CLINICAL TRIAL: NCT06771674
Title: Real-world Study of Patients With Human Papillomavirus-positive Recurrent/ Metastatic Oropharyngeal Squamous Cell Carcinoma Treated With First Line Pembrolizumab or Nivolumab With or Without Chemotherapy
Brief Title: Real-world Study of First Line Pembrolizumab- or Nivolumab-treated HPV-positive Recurrent/Metastatic Oropharyngeal Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Hookipa Biotech GmbH (Industry)
Collaborators: Cardinal Health (Industry)
Responsible Party: Sponsor
Other Study IDs: H-RWE-001
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma
Keywords: oropharyngeal squamous cell carcinoma; throat; head and neck cancer; squamous cell cancer; OPSCC; HNSCC; human papillomavirus; HPV; immunotherapy; real-world study; PD-L1 therapy; checkpoint inhibitor; pembrolizumab; nivolumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Neoplasms, Squamous Cell | interventions — pembrolizumab; Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- ECA 1: A representative sample of real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab monotherapy.
  Interventions: Drug: Pembrolizumab
- ECA 3: A representative sample of real-world patients with HPV+ R/M OPSCC and high CPS (at least 20 or more) treated with 1L pembrolizumab monotherapy.
  Interventions: Drug: Pembrolizumab
- ECA 2: A representative sample of real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab or nivolumab with chemotherapy.
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab
- ECA 4: A representative sample of real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab or nivolumab with or without chemotherapy.
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Given as monotherapy.
  Other Names: Keytruda
  Groups: ECA 1; ECA 3
Drug: Nivolumab — Given in combination with chemotherapy.
  Other Names: Opdivo
  Groups: ECA 2; ECA 4
Drug: Nivolumab — Given without chemotherapy.
  Other Names: Opdivo
  Groups: ECA 4
Drug: Pembrolizumab — Given in combination with chemotherapy.
  Other Names: Keytruda
  Groups: ECA 2; ECA 4
Drug: Pembrolizumab — Given without chemotherapy.
  Groups: ECA 4

SUMMARY:
Pembrolizumab and nivolumab (with or without chemotherapy) are used to treat head and neck cancer. The middle part of the throat (oropharynx) is a common location for head and neck cancer. This cancer is known as oropharyngeal squamous cell carcinoma (OPSCC) and is most often caused by human papillomavirus (HPV) infection. This real-world evidence study carried out in the United States (US) will assess patient demographic and clinical characteristics, treatment patterns, and effectiveness of pembrolizumab and nivolumab (with or without chemotherapy) in patients with HPV positive (HPV+) OPSCC after their cancer spread (metastatic) and/or returned (recurrent). The collected real-world data can be compared with data derived from matched study populations in clinical studies that test new therapies in patients with HPV+ OPSCC. This will allow a more reliable evaluation of the clinical benefits and better-informed design of future clinical studies in this patient population.

DETAILED DESCRIPTION:
This non-interventional study will be conducted as a single-phase, multicenter medical chart review of US patients with HPV+ recurrent and/or metastatic (R/M) OPSCC treated with first-line (1L) pembrolizumab or nivolumab (with or without chemotherapy). Participating physicians (Cardinal Health's Oncology Provider Extended Network) and clinical sites (Practice Research Network) will be asked to submit data on patient demographics, clinical characteristics, treatment patterns, and 1L treatment outcomes during a 10-week data collection period. The networks do not overlap, eliminating the chance of duplicate patient records. The completion of data collection defines the study completion date. The data collection period will be followed by a data validation period based on responses of the participating physicians and clinical sites to follow-up questions.

The data obtained in this study will create external control arms (ECAs) comprised of patients with HPV+ R/M OPSCC initiating 1L therapy with pembrolizumab monotherapy, or nivolumab with or without chemotherapy. The use of these ECAs will allow for a more accurate estimation of the effectiveness of therapies currently assessed in interventional clinical studies versus pembrolizumab or nivolumab (with or without chemotherapy) as assessed in this observational study in a non-randomized setting. This information will serve to increase the reliability of the study data from interventional clinical studies investigating therapies in matching indications and patient populations and improve the accuracy of the clinical data to inform future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HPV+ R/M OPSCC (base and posterior one-third of tongue, the tonsils, soft palate, and lateral pharyngeal walls).
* Initiated and treated with pembrolizumab monotherapy, or nivolumab (monotherapy or in combination with chemotherapy) as 1L therapy for HPV+ R/M OPSCC on or after 05 June 2024 (may have had curative intent treatment including surgery, chemotherapy, and/or radiotherapy for non-metastatic/non-recurrent disease).
* Have access to baseline assessment scan within 30 days prior to initiating 1L therapy for HPV+ R/M OPSCC and response assessment confirmed by objective measurements within 26 weeks of initiation of 1L therapy.
* Must have been followed for 6 months or more since initiation of 1L therapy for R/M OPSCC.

Exclusion Criteria:

* Participation in a controlled clinical trial for 1L R/M OPSCC.
* Central nervous system involvement or other concurrent malignancy at the time of 1L initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-world patients with HPV+ R/M OPSCC who received 1L pembrolizumab monotherapy, or nivolumab with or without chemotherapy will be evaluated. The ECAs derived from this real-world study are matched to respective study populations from interventional clinical studies. Propensity score matching will be used to generate the ECAs. The baseline characteristics used for matching will encompass key demographic and clinical factors potentially associated with treatment outcomes and may include:
  * Type of disease (only recurrent/metastatic including any recurrent)
  * Smoking history
  * Sex at birth
  * Race/Ethnicity
  * Hemoglobin
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Patient demographics with ECA 1 | Whole study period (05 June 2024 through 30 April 2025)
  Patient demographics among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab monotherapy.
Clinical characteristics with ECA 1 | Whole study period (05 June 2024 through 30 April 2025)
  Clinical characteristics among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab monotherapy.
Treatment patterns with ECA 1 | Whole study period (05 June 2024 through 30 April 2025)
  Treatment patterns among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab monotherapy.
1L treatment outcomes with ECA 1 | Whole study period (05 June 2024 through 30 April 2025)
  1L treatment outcomes among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab monotherapy.
Patient demographics with ECA 2 | Whole study period (05 June 2024 through 30 April 2025)
  Patient demographics among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab or nivolumab with chemotherapy.
Clinical characteristics with ECA 2 | Whole study period (05 June 2024 through 30 April 2025)
  Describe the clinical characteristics among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab or nivolumab with chemotherapy.
1L treatment outcomes with ECA 2 | Whole study period (05 June 2024 through 30 April 2025)
  1L treatment outcomes among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab or nivolumab with chemotherapy.
Treatment patterns with ECA 2 | Whole study period (05 June 2024 through 30 April 2025)
  Treatment patterns among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab or nivolumab with chemotherapy.
Patient demographics with ECA3 | Whole study period (05 June 2024 through 30 April 2025)
  Patient demographics among real-world patients with HPV+ R/M OPSCC and with a CPS of at least 20 or more treated with 1L pembrolizumab monotherapy.
Clinical characteristics with ECA3 | Whole study period (05 June 2024 through 30 April 2025)
  Clinical characteristics among real-world patients with HPV+ R/M OPSCC and with a CPS of at least 20 or more treated with 1L pembrolizumab monotherapy.
Treatment patterns with ECA3 | Whole study period (05 June 2024 through 30 April 2025)
  Treatment patterns among real-world patients with HPV+ R/M OPSCC and with a CPS of at least 20 or more treated with 1L pembrolizumab monotherapy.
1L treatment outcomes with ECA3 | Whole study period (05 June 2024 through 30 April 2025)
  1L treatment outcomes among real-world patients with HPV+ R/M OPSCC and with a CPS of at least 20 or more treated with 1L pembrolizumab monotherapy.
Patient demographics with ECA 4 | Whole study period (05 June 2024 through 30 April 2025)
  Patient demographics among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab or nivolumab with or without chemotherapy.
Clinical characteristics with ECA 4 | Whole study period (05 June 2024 through 30 April 2025)
  Describe the clinical characteristics among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab or nivolumab with or without chemotherapy.
Treatment patterns with ECA 4 | Whole study period (05 June 2024 through 30 April 2025)
  Treatment patterns among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab or nivolumab with or without chemotherapy.
1L treatment outcomes with ECA 4 | Whole study period (05 June 2024 through 30 April 2025)
  1L treatment outcomes among real-world patients with HPV+ R/M OPSCC treated with 1L pembrolizumab or nivolumab with or without chemotherapy.

SECONDARY OUTCOMES:
Real-world ECA 1 population versus a population from an interventional clinical study | Whole study period (05 June 2024 through 30 April 2025)
  Compare clinical outcomes of a matched patient population from an interventional clinical study with those of the representative ECA 1 real-world population with HPV+ R/M OPSCC treated with 1L pembrolizumab monotherapy from this study.
Real-world ECA 2 population versus a population from an interventional clinical study | Whole study period (05 June 2024 through 30 April 2025)
  Compare clinical outcomes of a matched patient population from an interventional clinical study with those of the representative ECA 2 real-world population with HPV+ R/M OPSCC treated with pembrolizumab or nivolumab with chemotherapy from this study.
Real-world ECA 3 population versus a population from an interventional clinical study | Whole study period (05 June 2024 through 30 April 2025)
  Compare clinical outcomes of a matched patient population from an interventional clinical study with those of the representative ECA 3 real-world population with HPV+ R/M OPSCC and with CPS of at least 20 or more treated with pembrolizumab monotherapy from this study.
Real-world ECA 4 population versus a population from an interventional clinical study | Whole study period (05 June 2024 through 30 April 2025)
  Compare clinical outcomes of a matched patient population from an interventional clinical study with those of the representative ECA 4 real-world population with HPV+ R/M OPSCC treated with pembrolizumab or nivolumab with or without chemotherapy from this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardinal Health, Dublin, Ohio, United States